CLINICAL TRIAL: NCT02503891
Title: Total Hip Replacement - MP-1 Acetabular Liner
Brief Title: AL-2 MP-1 (Polyimide) Acetabular Liner
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: M.M.A Tech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-01
Record Dates: First submitted 2015-07-14; First posted 2015-07-21 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis; Congenital Dysplasia of the Hip; Ankylosing Spondylitis; Post-traumatic; Arthrosis; Injury of Hip
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid; Hip Dislocation, Congenital; Spondylitis, Ankylosing; Hip Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Polymer on Ceramic (Experimental): MP-1 Polymer on Ceramic articulation system
  Interventions: Device: MP-1 Polymer on Ceramic Articulation system

INTERVENTIONS:
Device: MP-1 Polymer on Ceramic Articulation system — MP-1 Polymer liner on Ceramic head
  Other Names: AL-2 MP-1 Polyimide Acetabular liner

SUMMARY:
M.M.A.TECH Ltd. product is an Acetabular Liner Family produced of an advanced polyimide - MP-1™.

M.M.A.TECH Ltd. produces the Liners according to EN ISO 13485:2012 approved manufacturing process and supplies them to the customer.

The aim of this study is to evaluate, in the frame of PMCF, the safety and performance of using AL-X MP1 Polyimide Acetabular liners in Total Hip Replacement surgery by clinical following up of patients for a period of 2 years .

DETAILED DESCRIPTION:
The procedure involves removal of the diseased parts of the joint, that is the damaged cartilage and adjacent bone, and replacing them with artificial parts which closely resemble in structure and/or function the removed native parts.

The artificial parts fit onto the reshaped bone and are fixed either with bone cement (e.g., polymethylmethacrylate) and press fit of the part(cemented), or by self-anchorage with bone ingrowth to its porous surface(cementless).

The design of the artificial parts may include a stem, a keel or pegs, which fit onto the medullary canal of the bone or into a hole pre-prepared in the bone. An artificial part may fit loosely and be fixed with bone cement, press-fit for self- anchorage or include extendible anchors which are retracted upon placement and extended thereafter so as to secure the implant in place.

Following fixation of the components, the joint is reduced and the soft tissue tension is appropriately checked to reassure stability of the joint.

The MP-1™ acetabular liner will be tapper locked in acetabular metal shells to resurface the acetabular socket in cementless total hip replacement.

MMaTech Ltd will manufacture the liners to perfectly fit into the external metallic shell of the following sizes (mm):

LINER CUP SIZE LINER SIZE HEAD Liner thickness AL-2MP132040 44-48 32 ID 40 OD 32 4 mm AL-2MP136044 50-54 36 ID 44 OD 36 4mm AL-2MP136048 56-66 36 ID 48 OD 36 6mm AL-2MP140048 56-66 40 ID 48 OD 40 4mm

The MP-1™ Acteabular liners are intended to be used only against ceramic femoral heads- Biolox Delta

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for subject participation in the study are:

(Patient must meet all of the following characteristics to be enrolled in the study):

* Males and females, 21 to 90 years of age, inclusive;
* Primary diagnosis of non-inflammatory arthritis (osteoarthritis) or inflammatory arthritis (rheumatoid arthritis), or patients requiring a revision as specified previously;
* The patient or his/her legal guardian is willing to consent to participate in the study by signing and dating the approved consent form;
* The patient will be available for follow-up through at least two years postoperative;
* The patient has met an acceptable preoperative medical clearance and is free or treated for cardiac, pulmonary, hematological, etc., conditions that would pose excessive operative risk (FDA requirement);
* The patient has a total Harris Hip Score of less than or equal to 60 (FDA requirement);
* The patient meets none of the exclusion criteria.

Exclusion Criteria:

with any of the following characteristics must be excluded from the study):

* Patients known to have insufficient quantity or quality of bone support resulting from Conditions such as cancer, femoral osteotomy, Girdlestone resection, significant osteoporosis or metabolic disorders of calcified tissues. Patients with physical conditions tending to place extreme loads on implants such as morbid obesity (> 100 pounds over desirable body weight), Charcot joints, muscle deficiencies, or multiple joint disabilities;
* Patients with active localized or systemic infection;
* Patients who have not reached full skeletal maturity;
* Patient has had a total knee arthroplasty of either leg
* Patient psychological or neurological conditions which tend to preempt the patient's ability or willingness to restrict activities or follow medical advice, especially during the postoperative period, e.g.: drug or alcohol abuse, serious mental illness or retardation, or general neurological conditions;
* The patient is participating in any other pharmaceutical, biologic or medical device clinical investigation;
* Immunosuppressive disorders - immunosuppressive disorders are chronic conditions characterized by markedly inhibited ability to respond to antigenic stimuli. Examples of such conditions include patients who are on immunosuppressive therapy (corticosteroid hormones in large amounts, cytotoxic drugs, antilymphocytic serum or irradiation in large doses), patients receiving therapy to prevent homograft rejection, patients who have acquired immunodeficiency syndrome (AIDS), or auto-immune diseases (except rheumatoid arthritis).
* Pregnancy.
* Patients with known sensitivity to materials in the device.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Clinical patient status according to Harris Score | 6 months
  >60
Radiographic success | 3 mth , 12mth, 24 mth post-surgery
  o Radiographic success will be determined by femoral subsidence < 2mm, acetabular migration < 2mm, cup inclination < 4°, no acetabular or femoral osteolysis, and acetabular and femoral lucencies less than 50% of visible porous coating

CONTACTS AND LOCATIONS:
Overall Officials: Simha Sibony, Study Chair — M.M.A Tech Ltd.
Locations (1):
- Rambam Hospital, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
mmatech website